CLINICAL TRIAL: NCT06081374
Title: Determining the Effect of Simulation-based Breastfeeding Education on Breastfeeding Self-efficacy and Breastfeeding Problems: A Randomized Controlled Study
Brief Title: The Effect of Simulation-based Breastfeeding Education on Breastfeeding Self-efficacy and Breastfeeding Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, seda karaçay yıkar, Assistant professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 123
Record Dates: First submitted 2023-07-10; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-09

CONDITIONS: Postpartum Complication; Caesarean Section;Stillbirth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- simulation intervention (Experimental): simulation will be implemented.
  Interventions: Device: simulation implication
- education implication (Active Comparator): education will be implemented.
  Interventions: Device: simulation implication
- control group (No Intervention): no intervention will be made.

INTERVENTIONS:
Device: simulation implication — Breastfeeding education is planned by dressing pregnant women with simulation models.
  Other Names: nursing education
  Arms: education implication; simulation intervention

SUMMARY:
In the literature, there are studies conducted to determine the effect of simulation-based and different training techniques models given in the prenatal period on postpartum breastfeeding self-efficacy. However, no study was found that evaluated the effects of simulation-based and different training techniques given in the prenatal period on breastfeeding self-efficacy and breastfeeding problems. Therefore, this study was planned to determine the effect of simulation-based breastfeeding education on breastfeeding self-efficacy and breastfeeding problems in the prenatal period.

ELIGIBILITY:
Inclusion Criteria:

* Pregnants between32nd-36th gestational weeks,
* Primigravida,
* Planning to breastfeed,
* Can speak and understand Turkish,
* Pregnant women who agreed to participate in the study were included.

Exclusion Criteria:

* Breastfeeding contraindications,

  * Having a risky pregnancy, Having received a planned breastfeeding training before,
  * Premature birth (before 37th weeks of gestation),
* Having a systemic/chronic disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women will be included
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-11-01 (Estimated)

PRIMARY OUTCOMES:
simulation affect on breastfeeding self-efficacy | postpartum 7th week
  It is planned to increase women's breastfeeding self-efficacy through training Breastfeeding Self-efficacy scale points are supposed to be between 14-70 points. Getting higher points shows better breastfeeding self-efficacy.
simulation affect on breastfeeding problems | postpartum 7th week
  It is planned to prevent possible breast problems with the training given to women. It is supposed to get points from 18 to 90 related to Breastfeeding Experience Scale.Getting lower points is more preferable than higher points. Getting points near to 90 shows increased problems related to breastfeeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Seda Karaçay Yıkar, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
data will be kept in confident